CLINICAL TRIAL: NCT02194933
Title: Protocol 331-13-009: An Exploratory, Multicenter, Randomized, Double-Blind, fMRI Study of Fixed-dose Brexpiprazole (OPC-34712) (2 and 4 mg/Day Tablets) in Adults With Schizophrenia With Impulsivity
Brief Title: Monotherapy Brexpiprazole (OPC-34712) Trial in the Treatment of Adults With Schizophrenia With Impulsivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-13-009
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia With Impulsivity
Keywords: Schizophrenia; Mental Disorders, Antipsychotic,; Psychotic disorder, Impulsivity
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Impulsive Behavior | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brexpiprazole 2 mg (Experimental): Brexpiprazole 2 mg/day, once daily dose, tablet, orally
  Interventions: Drug: Brexpiprazole
- Brexpiprazole 4 mg (Experimental): Brexpiprazole 4 mg/day, once daily dose, tablet, orally
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole 2 mg/day, once daily dose, tablet, orally, for 6 weeks - Brexpiprazole 4 mg/day, once daily dose, tablet, orally, for 6 weeks
  Other Names: OPC-34712

SUMMARY:
The purpose of this study is to evaluate the effect of brexpiprazole, via functional magnetic resonance imaging (fMRI), on the right ventrolateral prefrontal cortex (VLPFC) activated by impulsive behavior.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 65 years of age, inclusive, at the time of informed consent (outpatients only), with a diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria and confirmed by both the M.I.N.I. for Schizophrenia and Psychotic Disorders Studies, and an adequate clinical psychiatric evaluation.
* Have a CGI-S score of ≤ 4 (moderately ill) at screening and baseline.
* Have a score of ≤ 4 (moderate) on PANSS item G8 (uncooperativeness) at screening and baseline.
* Have a BIS-11 score of ≥ 50 at screening and baseline.
* Willing to discontinue all prohibited psychotropic medications to meet protocol-required washouts prior to and during the trial period.
* Are stable on their current oral antipsychotic medication (no changes within the last month) and are able to meet protocol-required washouts of their current antipsychotic medication.
* Have received previous outpatient antipsychotic treatment at an adequate dose (at least minimal recommended dose for the treatment of schizophrenia according to the manufacturer labeling) for an adequate duration (at least 6 weeks) and showed a previous good response to such antipsychotic treatment (other than clozapine) in the last 12 months, according to the investigator's opinion.
* Subjects with eyesight that is sufficient to be able to see visual displays, or correctable with magnet-compatible glasses or contact lenses.
* Subjects fluent in English

Exclusion Criteria:

* Are presenting with schizophreniform or with a first episode of schizophrenia based on the clinical judgment of the investigator.
* Have been hospitalized for psychotic symptoms within the previous 6 months.
* Have a current DSM-IV-TR Axis I primary diagnosis other than schizophrenia, including, but not limited to, schizoaffective disorder, major depressive disorder, bipolar disorder, post-traumatic stress disorder, obsessive-compulsive disorder (OCD) or panic disorder, delirium, dementia, amnestic, or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, antisocial personality disorders, or mental retardation.
* Have worsening of ≥ 20% in total PANSS score between the screening and baseline assessments.
* Experiencing a deterioration in clinical status or an acute exacerbation of schizophrenia in the opinion of the Investigator.
* Experiencing acute onset of clinically significant depressive symptoms within the past 30 days, according to the investigator's opinion.
* Answer "Yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 6 months OR Answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR who, in the opinion of the investigator, present a serious risk of suicide.
* Have a history of stroke.
* Contraindications to magnetic resonance imaging (MRI) such as metal prostheses, pacemakers, claustrophobia, movement disorders, waist circumference more than 56 inches or head circumference more than 29 inches, color blindness, significant tremors, or history of head injury or prolonged unconsciousness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California at Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Derived] van Erp TG, Baker RA, Cox K, Okame T, Kojima Y, Eramo A, Potkin SG. Effect of brexpiprazole on control of impulsivity in schizophrenia: A randomized functional magnetic resonance imaging study. Psychiatry Res Neuroimaging. 2020 Jul 30;301:111085. doi: 10.1016/j.pscychresns.2020.111085. Epub 2020 May 5. PMID 32450497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States (US). 38 participants with schizophrenia with impulsivity were enrolled (signed informed consent) and randomized (1:1): 19 participants to brexpiprazole 2mg and 4mg treatment each; received at least 1 dose of Investigational medicinal product (IMP) for 6-week treatment phase in a double-blind design.
Pre-assignment Details: Participants had pretreatment screening phase from 2 to 21 days to assess eligibility criteria, complete screening assessments & to wash out from prior antipsychotic drugs & any other prohibited concomitant drugs; participants were followed for safety by clinic visits/telephone (after first 3 to 4 days of antipsychotic washout & weekly as needed).
Groups:
- Brexpiprazole 2 mg: Participants received Brexpiprazole 1 mg orally per day for 4 days followed by 2 mg per day until week 6 (Day 42)/early termination (ET)
- Brexpiprazole 4 mg: Participants received brexpiprazole 1 mg orally per day for 4 days followed by 2 mg per day for 3 days, 3 mg per day for 7 days and 4 mg per day until week 6 (Day 42)/ET.
Period: Overall Study
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Started | 19 | 19
Completed | 16 | 10
Not Completed | 3 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Participant met withdrawal criteria | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (10.0) | 47.4 (11.1) | 46.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Race [Number; unit: participants] — Different races were involved in this study
  participants
    Caucasian (White) | 6 | 7 | 13
    Black or African or American | 8 | 12 | 20
    Asian | 2 | 0 | 2
    Others | 3 | 0 | 3
Ethinicity [Number; unit: participants]
  Hispanic/Latino | 4 | 3 | 7
  Not Hispanic/Latino | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Brain Activation in the Ventrolateral Prefrontal Cortex (VLPFC) Based on Change From Baseline to Week 6 in fMRI Blood Oxygen-level Dependent (BOLD) Activation Score in the Right VLPFC During Performance of the Go/No-go Task
Description: To evaluate the effect of brexpiprazole on brain regions activated by impulsive behavior (specifically, activation of the right VLPFC). Assessed by fMRI measurements taken when participants perform tasks designed to assess impulsivity. The tasks to be performed in the scanner included the Go/No-go. Participants were asked to press a button as fast as they could to Stimulus A (eg, neutral face) that appeared on the screen (Go trials) & to NOT press a button to Stimulus B (eg, happy face) that appeared on the screen (No-go trials). The Go trials were presented at a higher frequency (eg, 75% of the time) than the No-go trials to build up a pre-potent response/response bias. Scores were not bounded by a minimum or maximum range, higher fMRI BOLD activation scores indicate increased brain blood flow, which reflects brain activity.
Time Frame: At baseline (Day 0), and week 6 (Day 42) of the treatment phase
Population: All participants who had a valid baseline and a Week 6 fMRI scan assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale
  At Week 0: number analyzed (Participants) | 14 | 13
  At Week 0 | 0.06450 (0.02815) | 0.06609 (0.02875)
  At Week 6: number analyzed (Participants) | 13 | 10
  At Week 6 | 0.04949 (0.02878) | 0.04326 (0.03128)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.3992, Mixed Models Analysis — Test for Baseline vs. Week 6

2. Primary Outcome: Change From Baseline Brain Activation in the VLPFC Based on Change From Baseline to Week 6 in fMRI BOLD Activation Score in the Right VLPFC During Performance of the SSRT Task
Description: To evaluate the effect of brexpiprazole on brain regions activated by impulsive behavior (specifically, activation of the right VLPFC). Assessed by fMRI measurements taken when participants performed impulsivity assessment tasks. A white circle was shown for 500ms, followed by a left (<)/right (>) arrow. When an arrow was presented, participants responded as fast as possible with their index/middle finger. A titration procedure with 4 staircases started with stop signal delay (SSD) values of 100, 150, 200 & 250ms to determine participant's SSRT. The tasks included 3 runs with 166 repetition times (TRs), TR=2s; 5 minutes, 32 seconds/run; 96 go trials, 32 stop trials/ run. The total task duration was 16 minutes & 36 seconds. Scores were not bounded by a minimum or maximum range, higher fMRI BOLD activation scores indicate increased brain blood flow, which reflects brain activity.
Time Frame: At baseline (Day 0), and week 6 (Day 42) of the treatment phase
Population: All participants who had a valid baseline and a valid Week 3 or Week 6 fMRI scan assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale
  At Week 0: number analyzed (Participants) | 15 | 14
  At Week 0 | 0.05200 (0.02993) | 0.09485 (0.03428)
  At Week 6: number analyzed (Participants) | 11 | 10
  At Week 6 | -0.00140 (0.03048) | 0.002815 (0.03541)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis — Test for Baseline vs. Week 6

3. Secondary Outcome: Change From Baseline to Week 3 in fMRI BOLD Activation Score in the Right VLPFC, Scanned by fMRI During Performance of Tasks Associated With Impulsivity (SSRT Task, Go/No-go Task)
Description: Go/No-go: Participants were to press button fast to Stimulus A (neutral face) (Go trials) & to NOT press button to Stimulus B (happy face) (No-go trials). Task comprised 4 runs of 3 minutes & 8 seconds each. Each run included 36 target (Go) & 13 non target (No-go) stimuli. The stimuli were presented for 500ms with 2 to 14.5 inter-stimulus interval fixation cross in between. Target stimuli were pseudo-randomized across runs so that each participant was presented with 2 Happy Go & 2 Neutral Go conditions.
  SSRT: White circle was shown for 500ms, followed by left (<)/right (>) arrow. When an arrow was presented, participants were to respond fast with their index/middle finger. A titration procedure with 4 staircases that started with stop signal delay (SSD) values of 100, 150, 200 & 250ms determined participant's SSRT.
  Scores were not bounded by a minimum or maximum range, higher fMRI BOLD activation scores indicate increased brain blood flow, which reflects brain activity.
Time Frame: At baseline (Day 0), and week 3 (Day 21) of the treatment phase
Population: All participants who had a valid baseline and a valid Week 3 fMRI scan assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale
  GNG; Week 0: number analyzed (Participants) | 14 | 13
  GNG; Week 0 | 0.06347 (0.02801) | 0.06553 (0.02869)
  GNG; Week 3: number analyzed (Participants) | 14 | 13
  GNG; Week 3 | 0.08523 (0.02801) | 0.04973 (0.02869)
  SSRT; Week 0: number analyzed (Participants) | 15 | 11
  SSRT; Week 0 | 0.05376 (0.02903) | 0.09550 (0.03346)
  SSRT; Week 3: number analyzed (Participants) | 14 | 11
  SSRT; Week 3 | 0.06398 (0.02979) | 0.02410 (0.03346)

4. Secondary Outcome: Change From Baseline to Week 6 in Barratt Impulsiveness Scale (BIS-11)
Description: A participant-rated scale was used to assess impulsive personality traits. The BIS-11 consisted of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/ always) and the scores were used to assess 6 first-order factors (attention, motor, self-control, cognitive complexity, perseverance and cognitive instability impulsiveness) and 3 second-order factors ( motor impulsiveness, nonplanning impulsiveness and attentional impulsiveness). The total score ranged from 30 to 120 with higher scores indicating impulsive personality traits, and took 10 to 15 minutes to complete the BIS-11.
Time Frame: At baseline (Day 0), and Week 6 (Day 42) of the treatment.
Population: The full analysis set consisted of all participants who took at least one dose of brexpiprazole and who had a valid baseline assessment and at least one valid postbaseline efficacy assessment. Change from baseline data were presented for participant count of 16, 12 for 2mg and 4mg arms, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 16 | 12
units on a scale | -2.6 (1.8) | 1.0 (2.0)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.1559, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.6201, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline to Week 3 in BIS-11
Description: as for outcome 4
Time Frame: At baseline (Day 0), and Week 3 (Day 21) of the treatment.
Population: All participants who took at least one dose of brexpiprazole and who had a valid baseline assessment and at least one valid postbaseline efficacy assessment. All participants who had a valid baseline and a valid Week 3 or Week 6 fMRI scan assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 16
units on a scale | -2.4 (1.7) | -2.3 (1.7)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.1642, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.1873, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline to Week 6 in Go/No-go Task Behavior
Description: Brexpiprazole reduced impulsivity was measured by a change in false alarm rate on the Go/No-go task (a lower false alarm rate was suggestive of better inhibition). Participants were instructed to press a button as fast as they could to Stimulus A (eg, neutral face) that appeared on the screen (Go trials) and to NOT press a button to Stimulus B (eg, happy face) that appeared on the screen (No-go trials). The stimuli were presented randomly. The value calculated was the rate of incorrect response for each condition (Go and No-go).
Time Frame: At baseline (Day 0), week 6 (Day 42) of the treatment phase
Population: All participants who took at least one dose of brexpiprazole and who had a valid baseline assessment and at least one valid postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
Millisecond
  At Week 0: number analyzed (Participants) | 14 | 13
  At Week 0 | 0.11 (0.08) | 0.09 (0.06)
  At Week 6: number analyzed (Participants) | 13 | 10
  At Week 6 | 0.08 (0.09) | 0.12 (0.17)

7. Secondary Outcome: Change From Baseline to Week 3 in Go/No-go Task Behavior
Description: as for outcome 6
Time Frame: At baseline (Day 0), and week 3 (Day 21) of the treatment phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
Millisecond
  Week 0: number analyzed (Participants) | 14 | 13
  Week 0 | 0.11 (0.08) | 0.09 (0.06)
  Week 3: number analyzed (Participants) | 14 | 13
  Week 3 | 0.10 (0.13) | 0.15 (0.14)

8. Secondary Outcome: Change From Baseline to Week 6 in Monetary Choice Questionnaire (MCQ) Score
Description: To measure "delay discounting" as an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The propensity of participants to delay reward was assessed with an MCQ. Discounting rate is estimated using, k= (A/V)1/D, where k is the discounting rate parameter, V is the immediate reward, A is the higher delayed reward and D is the amount of days to the delayed reward. The MCQ consisted of 27 choices between immediate and delayed rewards. The participants chose repeatedly between 2 hypothetical sums of money: a smaller amount now or a larger amount in the future (ex: ''Would you prefer $27 today or $50 in 21 days?"). The answers provided an estimate of the participant's discounting rate. The discounting rate parameter takes values between 0 and 1 and higher discounting rates indicated impulsivity. It took 5 to10 minutes to complete the MCQ
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale | -0.019762 (0.015213) | 0.023685 (0.017103)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.2061, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.1778, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline to Week 3 in MCQ Score
Description: To measure "delay discounting" as an index of impulsive behavior. It measured the extent to which the value of a reward decreased as the delay to obtaining that reward increased. The propensity of participants to delay reward was assessed with an MCQ. Discounting rate is estimated using, k= (A/V)1/D, where k is the discounting rate parameter, V is the immediate reward, A is the higher delayed reward and D is the amount of days to the delayed reward. The MCQ consisted of 27 choices between immediate and delayed rewards. The participants chose repeatedly between 2 hypothetical sums of money: a smaller amount now or a larger amount in the future (ex: ''Would you prefer $27 today or $50 in 21 days?"). The answers provided an estimate of the participant's discounting rate. The discounting rate parameter takes values between 0 and 1 and higher discounting rates indicated impulsivity.
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale | -0.012073 (0.014558) | 0.014520 (0.014891)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.4138, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.3375, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline to Week 6 in Stop Signal Reaction Time Task (SSRT) Task Behavior
Description: Brexpiprazole reduced impulsivity was measured by a change in Stop Signal Reaction Time (SSRT) on the SSRT task (a lower SSRT was suggestive of better inhibition). A white circle was shown for 500ms, followed by a left (<)/right (>) arrow. When an arrow was presented, participants responded as fast as possible with their index/middle finger. A titration procedure with 4 staircases started with stop signal delay (SSD) values of 100, 150, 200 & 250ms to determine participant's SSRT. The tasks included 3 runs with 166 repetition times (TRs), TR=2s; 5 minutes, 32 seconds/run; 96 go trials, 32 stop trials/ run. The total task duration was 16 minutes & 36 seconds. During scanning, the SSD was dynamically adjusted to yield a 50% successful inhibition rate, so that SSRT could be estimated for each participant. This resulted in approximately equal proportions of stop trials with & without a response
Time Frame: At baseline (Day 0), and Week 6 (Day 42).
Population: All participants who had a valid baseline and a valid Week 6 fMRI scan assessment
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
Millisecond
  At Week 0: number analyzed (Participants) | 12 | 10
  At Week 0 | 357.63 (61.51) | 323.25 (56.59)
  At Week 6: number analyzed (Participants) | 11 | 7
  At Week 6 | 299.68 (67.77) | 302.57 (34.68)

11. Secondary Outcome: Change From Baseline to Week 3 in SSRT Task Behavior
Description: as for outcome 10
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: All participants who had a valid baseline and a valid Week 3 fMRI scan assessment
Measure: Median (Standard Deviation); unit: Millisecond
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
Millisecond
  At week 0: number analyzed (Participants) | 12 | 10
  At week 0 | 357.63 (61.51) | 323.25 (56.59)
  At week 3: number analyzed (Participants) | 13 | 10
  At week 3 | 337.62 (76.23) | 328.05 (54.62)

12. Secondary Outcome: Change From Baseline to Week 6 in Continuous Performance Task (CPT) Behavior
Description: The AX trials were "target trials" with a valid cue followed by a valid probe X. This feature was intended to encourage participants to "expect" a valid probe to follow a valid cue. A consequence of this manipulation was that participants developed a prepotency to respond with "target" responses on trials for which valid cues were presented. The cue was presented for 1000msec, the inter-stimulus interval was 2000msec, and the target was presented for 500msec with a response window of 1500msec. The ITI was 1200msec. Participants had to practice until criteria were obtained. In the AX-CPT task, the subjects were instructed to press the "Yes" button every time there is a blue letter 'X' (target) following a white letter 'A' (cue). During this task, any letter appears on the screen randomly. The value calculated was the rate of correct response for all the reaction of target trial.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Rate of correct response
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
Rate of correct response | -0.70 (3.50) | -0.87 (4.06)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.8437, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.8318, Mixed Models Analysis

13. Secondary Outcome: Change From Baseline to Week 3 in CPT Behavior
Description: as for outcome 12
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Rate of correct response
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 14 | 14
Rate of correct response | 1.79 (4.14) | -0.61 (4.08)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.6697, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.8829, Mixed Models Analysis

14. Secondary Outcome: Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of 3 subscales containing 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. PANSS Positive and Negative subscale scores symptom constructs consisted of positive subscale (7 positive symptom constructs), negative subscale (7 negative symptom constructs), and general psychopathology subscale (16 symptom constructs). The possible maximum PANSS total score was 210; 30 indicating no symptoms; 210 indicating extremely severe symptoms.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 16 | 12
units on a scale | -2.4 (1.9) | -4.1 (2.1)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.2301, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.0599, Mixed Models Analysis

15. Secondary Outcome: Change From Baseline to Week 3 in PANSS Total Score
Description: as for outcome 14
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 16
units on a scale | -2.0 (1.4) | -2.3 (1.4)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.1595, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.1211, Mixed Models Analysis

16. Secondary Outcome: Change From Baseline to Week 6 in PANSS Positive Subscale Score
Description: PANSS consisted of positive subscales with 7 symptom constructs (delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility). Each item was scored using a scale of 1 to 7 (a higher score indicated increased severity). The maximum subscale score was 49; 7 indicated no symptoms; 49 indicated extreme severity.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 16 | 12
units on a scale | -1.4 (0.9) | -1.3 (1.0)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.1322, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.2113, Mixed Models Analysis

17. Secondary Outcome: Change From Baseline to Week 3 in PANSS Positive Subscale Score
Description: as for outcome 16
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 16
units on a scale | -1.2 (0.6) | -1.3 (0.6)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.0578, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.0588, Mixed Models Analysis

18. Secondary Outcome: Change From Baseline to Week 6 in PANSS Negative Subscale Score
Description: PANSS consisted of negative subscale with 7 symptom constructs (blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking). Each item was scored using a scale of 1 to 7 (a higher score indicated increased severity). The maximum subscale score was 49; 7 indicated no symptoms; 49 indicated extreme severity.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 16 | 12
units on a scale | -0.9 (0.6) | 0.2 (0.6)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.1666, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.7670, Mixed Models Analysis

19. Secondary Outcome: Change From Baseline to Week 3 in PANSS Negative Subscale Score
Description: as for outcome 18
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 16
units on a scale | 0.2 (0.7) | 0.8 (0.7)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.7178, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.2336, Mixed Models Analysis

20. Secondary Outcome: Change From Baseline to Week 6 in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score
Description: The severity of illness for each participant was assessed. The rater or investigator's response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 16 | 12
units on a scale | -0.1 (0.1) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.6558, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.9058, Mixed Models Analysis

21. Secondary Outcome: Change From Baseline to Week 3 in CGI-S Score
Description: as for outcome 20
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 16
units on a scale | -0.3 (0.1) | -0.1 (0.1)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg; Test type: Superiority or Other; p = 0.0078, Mixed Models Analysis
Statistical Analysis 2: Comparison: Brexpiprazole 4 mg; Test type: Superiority or Other; p = 0.4272, Mixed Models Analysis

22. Secondary Outcome: Clinical Global Impression - Improvement Scale (CGI-I) Score at Week 6
Description: To assess whether the total improvement was entirely due to drug treatment. The rater or investigator's response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The response at a given week was compared to the participant's condition at baseline (last available measurement at the baseline/Day 0 visit before the first dose of IMP).
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale | 3.6 (1.0) | 3.9 (0.5)

23. Secondary Outcome: CGI-I Score at Week 3
Description: as for outcome 22
Time Frame: During trial visits from Day 0 to Week 3 (Day 21).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 19 | 19
units on a scale | 3.7 (0.8) | 3.8 (0.5)

24. Secondary Outcome: Change From Baseline to Week 6 in Personal and Social Performance Scale (PSP)
Description: A validated clinician-rated scale that measured personal and social functioning in 4 domains: socially useful activities (eg, work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment was rated as absent, mild, manifest, marked, severe, or very severe and were converted to a total score on a 100-point scale: 71 to 100 - mild functional difficulty, 31 to 70 - manifest disabilities of various degrees and 1 to 30 - minimal functioning that required intense support and/or supervision.
Time Frame: During trial visits from Day 0 to Week 6 (Day 42).
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 17 | 14
units on a scale | 1.7 (1.6) | -0.0 (1.7)

ADVERSE EVENTS:
Time Frame: Trial visits (Days 0 to 42)
Description: An adverse event (AE) was any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug-related. Suspected adverse reaction (AR) - any AE caused by drug; in drug safety reporting, "reasonable possibility" meant to suggest a causal relationship between the drug and the AE. A serious AE (SAE) included any event that resulted in death, life-threatening, inability, hospitalization, congenital anomaly and requirement of medical/surgical intervention
Arm/Group | Brexpiprazole 2 mg | Brexpiprazole 4 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 13/19 | 14/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2 mg (N=19) | Brexpiprazole 4 mg (N=19)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Akathisia (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 2
Somnolence (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Irritability (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less